CLINICAL TRIAL: NCT06873334
Title: A Phase 2/3 Randomized, Double Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Pharmacodynamics, Safety and Efficacy of SKY-0515 in Participants With Huntington's Disease
Brief Title: Study of SKY-0515 for Safety, Efficacy, and Pharmacodynamics in Participants With Huntington's Disease
Acronym: Falcon-HD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Skyhawk Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKY-0515-004-ANZ
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Huntington Disease; Huntingtons Disease
Keywords: Sky-0515; Skyhawk; Mutant Huntington protein; HTT; mRNA; Huntington Disease; Splicing; Huntingtons Disease; Neurodegenerative
MeSH Terms: conditions — Huntington Disease; Chorea

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled dose ranging.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 (Active) (Active Comparator): Dosage Level(s): Low dose once daily oral
  Interventions: Drug: SKY-0515
- 2 (Active) (Active Comparator): Dosage Level(s): Mid dose once daily oral
  Interventions: Drug: SKY-0515
- 3 (Active) (Active Comparator): Dosage Level(s): High dose once daily oral
  Interventions: Drug: SKY-0515
- 4 (Control) (Placebo Comparator): Matching placebo once daily oral
  Interventions: Drug: SKY-0515 Placebo

INTERVENTIONS:
Drug: SKY-0515 — Study Drug Name (INN): SKY-0515 Type: Drug (small molecule) Dosage Level(s): Low, mid, high Route of Administration: Oral Dosage Frequency: Once daily Blinded Treatment Duration: 12 months
  Use: Experimental Sourcing: SKY-0515 will be provided centrally by the Sponsor or subsidiary, or designee Packaging and Labeling: Study drug will be provided in blinded bottles labeled as required per country requirement. All packaging and labeling operations for the study drug will be performed according to current Good Manufacturing Practice for Medicinal Products and the relevant regulatory requirements.
  Arms: 1 (Active); 2 (Active); 3 (Active)
Drug: SKY-0515 Placebo — Route of Administration: Oral Dosage
  Frequency: Once daily
  Blinded Treatment Duration: 12 months
  Use: Experimental
  Sourcing: SKY-0515 placebo will be provided centrally by the Sponsor or subsidiary, or designee
  Packaging and Labeling: Study drug will be provided in blinded bottles labeled as required per country requirement. All packaging and labeling operations for the study drug will be performed according to current Good Manufacturing Practice for Medicinal Products and the relevant regulatory requirements
  Arms: 4 (Control)

SUMMARY:
The goal of this clinical trial is to test if the drug SKY-0515, an oral medication, can lower harmful proteins linked to Huntington's Disease (HD) and improve the symptoms of participants with HD.

This study includes men and women aged 25 and older who have HD confirmed by genetic testing and meet certain requirements for physical ability and independence.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the safety, pharmacodynamics, and efficacy of SKY-0515, a novel, orally-administered small molecule mRNA-splicing modulator for treating Huntington's Disease (HD). HD is a rare, inherited neurodegenerative condition caused by a mutation in the huntingtin (HTT) gene, resulting in excessive production of mutant huntingtin (mHTT) protein, which damages nerve cells and leads to progressive motor, cognitive, and psychiatric symptoms.

SKY-0515 is designed to reduce mHTT protein levels by lowering of HTT messenger RNA (mRNA) through a splicing mechanism, leading to a decrease in both wild-type and mutant forms of HTT protein. Additionally, the drug lowers postmeiotic segregation 1 (PMS1) protein, which plays a role in somatic CAG repeat expansion-a key driver of HD progression. In early studies, SKY-0515 has reduced HTT and PMS1 mRNA levels in a dose-dependent manner, with favorable safety and tolerability profiles in healthy volunteers.

This study is a randomized, double-blind, placebo-controlled, trial conducted at multiple sites. Participants must be aged 25 or older, have genetically confirmed HD (CAG repeat length ≥ 40), and meet specific functional and motor criteria. They will be assigned randomly to one of four treatment arms (three doses of SKY-0515 and one placebo group) in a 1:1:1:1 ratio.

The study is composed of three periods:

1. Screening Period (up to 4 weeks): Participants will undergo eligibility assessments.
2. Double-Blind Treatment Period (12 months): Participants will take SKY-0515 or a placebo once daily and undergo regular clinic visits for monitoring. Safety and efficacy will be evaluated through blood tests, imaging (MRI), and clinical assessments, including the Unified Huntington's Disease Rating Scale (UHDRS).
3. Follow-Up Period (4 weeks): After completing treatment, participants will be monitored for any remaining effects.

An independent Data Safety Monitoring Board (DSMB) will oversee the trial to ensure participant safety.

This study will assess:

* Changes in levels of HTT proteins and other HD-related biomarkers.
* Effects on HD-related brain atrophy and clinical features.
* Long-term safety of SKY-0515.

ELIGIBILITY:
Inclusion Criteria:

* You must be 25 years or older.
* You must have Huntington's Disease confirmed through genetic testing, with a specific gene change (CAG repeat of 40 or more).
* Total Functional Capacity (TFC) score of 10 or more).
* Total Motor Score (TMS) of 6 or more).
* Independence Score (IS) of 70 or more).
* Women who can have children must have a negative pregnancy test before starting and use two types of birth control during the study and for 30 days after the last dose of the study drug.
* Men must agree to use birth control during the study and for 90 days after the last dose.
* You must agree to sign a consent form and follow the study's rules and schedule.

Exclusion Criteria:

* You have other serious health problems or brain/spinal issues that could interfere with the study or make procedures unsafe.
* You have a condition that interferes with protocol-specified assessments, like an implanted medical device or difficulty getting an MRI.
* You have cancer, except for some types of skin cancer, or a history of cancer in the last five years.
* You have severe allergies or have reacted badly to similar drugs in the past.
* You are taking medications or treatments that might interfere with the study.
* You've been in another study or taken experimental drugs in the last two months (or longer for some drugs).
* You have had any kind of gene therapy.
* You have a history of suicidal thoughts, severe depression, or have attempted suicide in the past year.
* Your liver function tests show significant abnormalities.
* You have tested positive for hepatitis B, hepatitis C, or HIV.
* You are pregnant, breastfeeding, or planning to become pregnant during the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in blood mHTT protein levels | 12 months
Changes in brain volume measured through MRI | 12 months
Changes in UHDRS | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Mokhtarani, MD, Study Director — Skyhawk Therapeutics, Inc.
Locations (11):
- Australia (7):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The University of Queensland, Herston, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - The Perron Institute for Neurology and Translational Science (Perron Institute), Nedlands, Western Australia
- New Zealand (4):
  - Huntington's Disease Association, Auckland
  - Auckland City Hospital, Auckland
  - Christchurch Neurology Trials Limited, Christchurch
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Skyhawk Therapeutics Website — https://www.skyhawktx.com/